CLINICAL TRIAL: NCT06007833
Title: The Investigation of the Effects of Physical Therapy and Rehabilitation Applications on the Hip and Defined Functional Parameters in Children With Developmental Hip Dysplasia
Brief Title: Physical Therapy Applications on the Hip and Defined Functional Parameters in Children With Developmental Hip Dysplasia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Elisa Çalışgan, The Investigation of the Effects of Physical Therapy and Rehabilitation Applications on the Hip and Defined Functional Parameters in Children with Developmental Hip Dysplasia, Inonu University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022/3832
Record Dates: First submitted 2023-08-10; First posted 2023-08-23 (Actual); Last update posted 2023-08-23 (Actual); Status verified 2023-08

CONDITIONS: Exercise; Developmental Dysplasia of the Hip
Keywords: Dysplasia; Hip subluxation; Dislocation; Rehabilitation
MeSH Terms: conditions — Motor Activity; Developmental Dysplasia of the Hip; Joint Dislocations | interventions — Physical Therapy Modalities

STUDY DESIGN:
Intervention Model Description: Experimental, Randomized Controlled Study
Who Masked: Participant
Masking Description: Participants didn't know taking which exercise treatment methods.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- physical therapy and rehabilitation program in addition to conservative treatment (Experimental): Orthoses and positioning will be applied to the experimental group as a conservative treatment, following post-surgical plastering. In addition, they will receive a physical therapy and rehabilitation program
  Interventions: Behavioral: Physical Therapy and Rehabilitation Modalities
- Conventional Group (Active Comparator): As a conservative treatment in the control group, post-surgical plastering followed by orthoses and positioning will be applied
  Interventions: Behavioral: Conventional Group

INTERVENTIONS:
Behavioral: Physical Therapy and Rehabilitation Modalities — In the experimental group, the subjects who were taken to the physical therapy modality in addition to conventional therapy. Total, each session was performed for 60 minutes, 8 weeks, 3 days a week, under the supervision of a physiotherapist, while the other days, the family member performed 3 times a day, each movement for 3 sets, 10-15 repetitions, for a total of 60 minutes. A rest interval of less than 2 minutes was given between each set. By making use of heat modalities before starting the exercises, the elongation ability of the warmed tense structure was increased and the risk of damage in stretching exercises was reduced. The cold application was applied to the soft tissues in the extended position for 1-2 minutes with a cold pack, as the application of cold immediately after the stretching would ensure the preservation of the range of motion. Progress in the exercise program; adjusted for strength, endurance, flexibility, balance and functionality parameters.
  Arms: physical therapy and rehabilitation program in addition to conservative treatment
Behavioral: Conventional Group — As a conservative treatment in the control group, post-surgical plastering followed by orthoses and positioning was applied.
  Arms: Conventional Group

SUMMARY:
The aim of this study was to investigate the effects of physical therapy and rehabilitation applications on the hip and defined functional parameters in children with developmental hip dysplasia.

DETAILED DESCRIPTION:
Developmental dysplasia of the hip (DDH) is one of the most important factors causing disability in childhood. DDH is the reason for 29% of all primary hip replacements under 60 years of age. The treatment of DDH, which is applied after an average of 12 months of age in infants, becomes difficult due to shortening of the extra-articular soft tissues, acetabular dysplasia, capsular restriction, and increased femoral anteversion. In the treatment of subluxation, dislocation and residual acetabular dysplasia, many pelvic iliac osteotomies are actively applied to increase joint stability and compatibility of the femur acetabulum. The treatment method and physical therapy to be applied in the treatment of DDH vary depending on the age and type of pathology. Therefore, osteotomies can be performed in isolation or in combination with open reduction of the hip and femoral osteotomies. The general opinion about the minimum patient age for iliac osteotomies (Dega osteotomy, Salter innominate) is that it can be done in children who are at walking age. With Dega osteotomy, anterior, lateral and mainly posterior deficiencies are eliminated by changing the acetabular inclination and structure and increasing the grip between the femoral head and the acetabulum.

In the literature, there are studies on the examination of various angular values of the hip (alpha, beta, coverage angle), various classification methods, and whether the postoperative follow-up of children who underwent open, closed reduction and osteotomy requires a reconstructive surgical procedure. No studies have been found on the strength of the hip muscles due to the application of surgical techniques in children with DDH who have weak hip, chorea and lower extremity muscles due to intrauterine and structural conditions. There are no studies on how the affected muscles affect the hip parameters and functional capacities of children with DDH. We think that hip muscle strength, femoral head and anteversion angle, acetabular index, hip adductor muscle tension are important in terms of hip stability and functionality in children aged 2-5 years. Due to the lack of studies in this field in the literature, this study; The aim of this study was to examine the effects of physical therapy and rehabilitation practices on hip and determined functional parameters in children with developmental dysplasia of the hip.

ELIGIBILITY:
Inclusion Criteria:

* 2-5 years old,
* Diagnosed with developmental hip dysplasia,
* Have not undergone any foot surgery,
* Not having any neurological or rheumatological disease,
* Having sufficient cooperation to understand and correctly apply the tests,
* Patients with informed consent from their families were included.

Exclusion Criteria:

* Having neurological problems,
* Meningomyelocele (diagnosed with Spina Bifida),
* Mental retardation and uncooperative,
* Children with inflammation, spasticity, spina bifida, arthrocentesis,
* Down syndrome-related dislocation,
* Children who could not obtain informed consent from their families were excluded from the study.

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2023-10-30 (Estimated); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
The Evaluation of Trunk Control | baseline and week 8
  Trunk Control Measurement Scale, This scale, which is applied to evaluate trunk control, consists of 2 sub-headings as static sitting balance and dynamic sitting balance. The trunk control measurement scale includes a total of 15 items evaluating trunk control in children. Individuals; without back support, feet are in full contact with the ground, and hips and knees are seated in 90º flexion. In the static sitting balance subgroup (items 1-5), the patient's performance in maintaining trunk stabilization while the upper and lower extremities are in motion is evaluated. It consists of dynamic sitting balance parameters (item 6-15), selective movement control (item 6-12) and dynamic reaching subscale (item 13-15). Functional reach, which is a sub-parameter of dynamic sitting balance, is an important parameter in evaluating balance in children. Scoring of this scale varies between 0-58; A higher score indicates better trunk control.

SECONDARY OUTCOMES:
The Evaluation of the Endurance of the Spinal Stability Muscles | baseline and week 8
  Modified "Biering-Sorensen" trunk extension, trunk flexion test, lateral and prone bridge test are applied to evaluate the static endurance of spinal stability muscles. The number of repetitions completed by the patients within a 30-second test interval is documented; a higher number of repetitions indicate strong performance.
The Evaluation of the Strength of the Spinal Stability Muscles | baseline and week 8
  "Sit-ups" and Modified "Push-ups" tests are applied to evaluate the strength of spinal stability muscles. The number of repetitions that the patients could do for 30 seconds during the test is recorded.
The Evaluation with Radiological Imaging of Hip Parameters | baseline and week 8
  Femoral head ossification in mm, femoral inclination angle in degrees, acetabular index developments in degrees will be examined.
The Assessment of Aerobic Capacity | baseline and week 8
  The 1-min walk test is used to evaluate the walking capacity of a pediatric individual, which is defined as the maximum walking speed.
The Evaluation of Anaerobic Capacity | baseline and week 8
  10m walking test is used to evaluate of anaerobic capacity. The time the child completes the 10-meter course at normal walking speed is recorded.
The Evaluation of the Dynamic Balance | baseline and week 8
  Timed get up and go test, evaluates the dynamic balance of individuals during functional mobility; It includes components such as standing, walking and turning. The children are asked to stand up without support from the chair they are sitting in, and to return from the designated area after walking a 3-meter distance at a normal pace and sit back in the chair without support. After a trial walk, the test is repeated three times; The average of the results is recorded. At the end of the test, the time calculated with the stopwatch is noted in seconds.
The Evaluation of Functional Mobility and Dynamic Balance | baseline and week 8
  It is a simple test applied to evaluate functional mobility and dynamic balance. The child, who is standing at a height of 20 cm by the child's leg length and 30 cm away on a 10-step ladder, is told to go up and down the stairs as quickly and safely as he can.
The Evaluation of Muscle Strength | baseline and week 8
  In muscle strength measurements; hip flexors, abductors, extensors, knee flexors and extensors, foot dorsiflexors and plantar flexors are evaluated. Manual Muscle Testing System (Lafayette Instrument Company, Lafayette, AB) (Lafeyette), an easy-to-carry, easy-to-use, inexpensive and portable handheld dynamometer, is used to measure maximum muscle strength for our measurements.

CONTACTS AND LOCATIONS:
Overall Officials: Elisa Calisgan, PhD, Principal Investigator — Inonu University
Locations (1):
- Inonu University, Malatya, Turkey (Türkiye)